CLINICAL TRIAL: NCT04842240
Title: Comparison of Patient Reported Outcome Measures in Patients Undergoing Pre Versus Sub-pectoral Implant Based Breast Reconstruction
Brief Title: Comparison of Patient Reported Outcome Measures Using the BREAST-Q Questionnaire in Patients Undergoing Pre Versus Sub-pectoral Implant Based Immediate Breast Reconstruction.
Acronym: PROM-Q
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 283017
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Breast Disease; Breast Cancer; Patient Satisfaction; Surgery
Keywords: Breast reconstruction; Breast implant; Patient reported outcome measures
MeSH Terms: conditions — Breast Diseases; Breast Neoplasms; Patient Satisfaction | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing implant based immediate breast reconstruction.: Patients will undergo either pre- or sub-pectoral implant based immediate breast reconstruction.
  Interventions: Procedure: Pre- or sub-pectoral implant based immediate breast reconstruction

INTERVENTIONS:
Procedure: Pre- or sub-pectoral implant based immediate breast reconstruction — All study participants will undergo skin sparing mastectomy (with or without nipple preservation) for breast cancer or for risk reduction. Patients will undergo immediate breast reconstruction using an implant or a tissue expander. The device will be placed in pre- or sub-pectoral plane which will be supported by mesh (Tiloop/Surgimend Acellular Dermal Matrix) and/or a dermal flap.

SUMMARY:
The PROM Q study aims to compare patient reported outcome measures (PROMs) in patients undergoing mastectomy and immediate implant based breast reconstruction (IBR). This is the commonest form of breast reconstruction and current advances in surgical technology have led to increasing number of patients having implants placed above the pectoral muscle (pre-pectoral), rather than below it (sub-pectoral). This has important benefits for patients including shorter surgery time, quicker recovery, and avoidance of animation deformity (visible muscle twitching of the reconstructed breast) as the pectoral muscle is not divided to cover the implant. However, potential disadvantages include rippling effect as the implant is covered by the skin and subcutaneous tissue only, as well as potentially higher risk of capsule (scar tissue) formation.

By utilising a validated questionnaire (BREAST-Q), we will assess for any difference in PROMs between the two groups of patients. The results will provide valuable information for future patients when making an informed decision about their reconstruction options. This questionnaire study will include consecutive patients undergoing mastectomy and immediate IBR for breast cancer as well as for risk reduction at Leeds Teaching Hospitals NHS Trust. The study participants will undergo either pre- or sub-pectoral IBR based on their informed discussion with the clinical team. This is a non-randomised observational study.

DETAILED DESCRIPTION:
Patients who undergo implant based immediate breast reconstruction (IBR) are offered an option of pre- versus sub-pectoral breast reconstruction. Both approaches are well established and have proven safety in terms of low rate of complication rates. However, we do not know if there is a significant difference in patient reported outcome measures (PROMs) between the two surgical techniques over time.

The study aims to investigate if the difference in the surgical technique for immediate implant breast reconstruction (pre- versus sub-pectoral) influences patient perceived outcomes. This is a prospective non-randomised longitudinal cohort study which will aim to recruit consecutive eligible patients undergoing mastectomy with immediate implant based reconstruction surgery for early breast cancer or risk reduction using repeated measures and mixed methods.

This study will utilise a well validated patient questionnaire for breast reconstruction (BREAST-Q; http://qportfolio.org/breast-q/breast-cancer/) and will be carried out at a teaching hospital breast unit. The specific objectives will be to compare aesthetic outcome, post-operative pain and functionality as reported by PROMs. The study participants will be followed up for 12 months. The PROMs data will be collected at baseline, 2 weeks, as well as at 3 and 12 months post-surgery. Matching data will be collected for each study participant including the type of surgery performed, patient characteristics, post-operative complications, and any recommended adjuvant treatment. These data will be correlated with the matching questionnaire results in order to explore for potential clinical factors which may influence PROMs.

ELIGIBILITY:
Inclusion Criteria:

* Skin or nipple sparing mastectomy with immediate implant based reconstruction for breast cancer or for risk reduction
* Unilateral or bilateral mastectomy
* Implant or expander based immediate reconstruction
* Able to read and understand questionnaire in English

Exclusion Criteria:

* Male or transgender
* Mastectomy only with no reconstruction
* Delayed reconstruction
* Autologous reconstruction
* Cognitive impairment or inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing mastectomy who opt to have immediate implant based reconstruction. This will be either patients undergoing breast cancer treatment or counselled with regards to risk reducing strategies for known germline breast cancer susceptibility gene mutations or at increased risk due to family history. The study will be carried out at a single teaching hospital breast unit.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To compare any difference in patient reported outcome measures in patients undergoing pre- versus sub-pectoral implant based breast reconstruction. | Up to 12 months post-surgery
  To measure the difference in BREAST-Q score in patients undergoing pre- versus sub-pectoral implant based breast reconstruction. We will compare psychosocial well-being, satisfaction with breasts, physical well-being, animation deformity, and patient experience with the clinical team.

CONTACTS AND LOCATIONS:
Overall Officials: Baek Kim, FRCS MD MA, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rampal R, Jones SJ, Hartup S, Robertson C, Tahir W, Jones SL, McKenzie S, Savage JA, Kim B. Three and twelve-month analysis of the PROM-Q study: comparison of patient-reported outcome measures using the BREAST-Q questionnaire in pre- vs. sub-pectoral implant-based immediate breast reconstruction. Breast Cancer Res Treat. 2024 Nov;208(2):275-282. doi: 10.1007/s10549-024-07416-5. Epub 2024 Jul 10. PMID 38985220

DOCUMENTS (1):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT04842240/Prot_000.pdf